CLINICAL TRIAL: NCT01050465
Title: MedlinePlus Health Prescriptions: Developing a Real World Approach for Clinic Use
Brief Title: MedlinePlus Health Prescriptions: Developing a Pragmatic Approach for Clinic Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HHSN276200800445P
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Acne Vulgaris; Allergic Rhinitis; Anxiety; Asthma; Back Pain; Prostatic Hyperplasia; Bursitis; Chronic Obstructive Pulmonary Disease; Cough; Coronary Artery Disease; Depression; Diabetes Mellitus; Diarrhea; Gastroesophageal Reflux; Fibromyalgia; Headache; HIV Infections; Hypothyroidism; Hyperlipidemia; Hypertension; Influenza; Sleep Initiation and Maintenance Disorders; Irritable Bowel Syndrome; Migraine Disorders; Obesity; Obstructive Sleep Apnea; Osteoarthritis; Senile Osteoporosis; Shoulder Pain; Sinusitis; Smoking Cessation; Tobacco Use Cessation; Menopause; Urinary Incontinence; Urinary Tract Infection; Vaginitis; Vertigo
Keywords: HIV; Knee pain; Colonoscopy; Mammography; Vaccination
MeSH Terms: conditions — Acne Vulgaris; Rhinitis, Allergic; Anxiety Disorders; Asthma; Back Pain; Prostatic Hyperplasia; Bursitis; Pulmonary Disease, Chronic Obstructive; Cough; Coronary Artery Disease; Depression; Diabetes Mellitus; Diarrhea; Gastroesophageal Reflux; Fibromyalgia; Headache; HIV Infections; Hypothyroidism; Hyperlipidemias; Hypertension; Influenza, Human; Sleep Initiation and Maintenance Disorders; Irritable Bowel Syndrome; Migraine Disorders; Obesity; Sleep Apnea, Obstructive; Osteoarthritis; Osteoporosis; Shoulder Pain; Sinusitis; Smoking Cessation; Tobacco Use Cessation; Urinary Incontinence; Urinary Tract Infections; Vaginitis; Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- email (Active Comparator): Patients randomized to this arm will receive an email health information prescription.
  Interventions: Other: health information prescription
- paper (Active Comparator): Patients randomized to this arm will receive a paper health information prescription.
  Interventions: Other: health information prescription

INTERVENTIONS:
Other: health information prescription — Patients randomized to the email arm will receive a health information prescription via email on a health care topic following their clinic visit. Patients randomized to the paper arm will receive a health information prescription on paper on a health care topic following their clinic visit.

SUMMARY:
The specific aim of this proposed pilot study is to compare two standardized processes (paper and electronic) to deliver a customized MedlinePlus health information prescription.

DETAILED DESCRIPTION:
The specific aim of this proposed pilot study is to compare two standardized processes (paper and electronic) to deliver a customized MedlinePlus health information prescription.

Primary Hypothesis. Individuals in the paper prescription group will be just as likely to seek information using MedlinePlus compared with individuals in the group who receive the same customized information through an email prescription.

Secondary Hypothesis. Individuals in the paper prescription group will be just as likely to have successful behavioral outcome measures as those in the group who receive the same customized information through an email prescription.

ELIGIBILITY:
Inclusion Criteria:

* one of the 40 target health conditions.

Exclusion Criteria

- absence of at least one of the target 40 conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 907 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
seeking information using MedlinePlus | clicks will be tracked on the website when they occur

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hodge, MD, Principal Investigator — University of Missouri-Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coberly E, Boren SA, Mittal M, Davis JW, Scoville C, Chitima-Matsiga R, Ge B, Cullina A, Logan RA, Steinmann WC, Hodge RH. MedlinePlus-based health information prescriptions: a comparison of email vs paper delivery. Inform Prim Care. 2012;20(3):197-205. doi: 10.14236/jhi.v20i3.25. PMID 23710844